CLINICAL TRIAL: NCT01921127
Title: A U.S. Retrospective Database Analysis Evaluating the Comparative Effectiveness of Budesonide/Formoterol (BFC) vs. Fluticasone/Salmeterol (FSC) Combination in Patients With COPD.
Brief Title: Comparative Effectiveness of Symbicort vs. Advair Among COPD Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 000152
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: COPD
Keywords: COPD, Comparative effectiveness, Symbicort
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Symbicort: BFC patients new to ICS/LABA therapies
- Advair: FSC patients new to ICS/LABA therapies.

SUMMARY:
This study is intended to evaluate treatment effectiveness of BFC compared to FSC in COPD patients new to ICS/LABA combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Continuous health plan enrollment for 12 months before and after index Rx, at least one prescription for BFC or FSC during intake period, naive to ICS/LABA therapies in year prior to first prescription claim, COPD diagnosis, aged 40 or over at time of first prescription.

Exclusion Criteria:

* ICS/LABA combination during pre-index period, patients with a claim for BFC and FSC on the same day, patients diagnosed with cancer, patients with long-term OCS medication use during pre-index period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health plan members with COPD aged 40 years or older receiving one or more prescriptions of BFC or FSC during 3/1/2009 and 3/31/2013 who are naive to ISC/LABA combinbination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rate of COPD exacerbation | 12 months
  The rate of COPD exacerbation will be defined as the total number of COPD exacerbations during the post-index period for all patients in each treatment cohort divided by the total number of person years. A COPD exacerbation event is defined as any of three conditions: COPD related inpatient hospitalization, COPD related emergency department visit, or COPD outpatient/office visit with a pharmacy claim for OCS and/or antibiotics on the same day or within ten days.

SECONDARY OUTCOMES:
COPD exacerbation rate sensitivity and subgroup analyses | 12 months
  The following sensitivity and subgroup analyses will be performed for the primary outcome: Time to first COPD exacerbation, on-treatment analysis, switchers and non-switchers.
COPD respiratory medication use | 12 months
  COPD respiratory medication, use for BFC and FSC will be described in post-index period by presenting total number of COPD medication classes filled. Antibiotic use will be assessed overall and within 10 days of OCS Rx.
COPD related healthcare utilization | 12 months
  COPD related outpatient/office visit, COPD related inpatient hospitalization length of stay, COPD related ICU admission and length of stay, COPD procedures.
All-cause utilization | 12 months
  Frequency of all-cause resource use of: inpatient hospitalizations and length of stay, ICU admissions and length of stay, and outpatient/office visits. Total number of different prescription medication classes filled will also be determined.
All- cause and COPD related healthcare costs | 12 months
  Costs will be reported for the following resource uses: inpatient hospitalizations, ED visits, outpatient/office visits, skilled nursing facility, total medical, and prescriptions. Costs will be reported for all-cause as well as COPD related.
Treatment patterns and adherence | 12 months
  Continuity of care during the 12 months post-index period will be measured with the Bice and Boxerman index. Proportion of Days Covered (PDC) and Medication Possession Ratio (MPR) will be used to measure the compliance of the index-medication (Symbicort or Advair).
Treatment modification | 12 months
  COPD medication use, such as treatment changes, will be captured post-index.
COPD exacerbation rate sensitivity analysis | up to 4 years
  All COPD exacerbation rates will be captured during the entire patient follow-up (beyond 12 months of the post index period) for BFC and FSC

OTHER OUTCOMES:
Pneumonia diagnosis validation | 12 months
  The diagnosis codes used to identify pneumonia in the claims database will be validated through medical chart review. For the validation analysis, the validity of claims will be evaluated by finding out whether or not the patient has a diagnosis of pneumonia in the claims.

REFERENCES:
- [Derived] Kern DM, Davis J, Williams SA, Tunceli O, Wu B, Hollis S, Strange C, Trudo F. Comparative effectiveness of budesonide/formoterol combination and fluticasone/salmeterol combination among chronic obstructive pulmonary disease patients new to controller treatment: a US administrative claims database study. Respir Res. 2015 Apr 23;16(1):52. doi: 10.1186/s12931-015-0210-x. PMID 25899176
- See also: Redacted protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1879&filename=AZN_COPD_Advair_CER_protocol_July_26_2013_FINAL_Redacted.pdf
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1879&filename=NCT01921127_SYM_Advair_Redacted.pdf